CLINICAL TRIAL: NCT05884216
Title: Entarik Feeding Tube System Placement in Adult ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on regulatory precedent for other smart feeding tubes, sufficient performance data was obtained to submit a 510(k) application with the FDA for the Entarik System.
Sponsor: Gravitas Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRD-04-1642-01
Record Dates: First submitted 2023-04-18; First posted 2023-06-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Nasogastric Tube

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Entarik (Experimental): Entarik FT System guided placement
  Interventions: Device: Entarik Feeding Tube System
- Control (Active Comparator): Entarik Ft placement placement not guided with monitor
  Interventions: Device: Entarik Feeding Tube System without monitoring

INTERVENTIONS:
Device: Entarik Feeding Tube System — Entarik Feeding Tube:
  The Entarik Feeding Tube is intended for the administration of nutrition, fluids and medications by the nasoenteric route for patients who have an intact gastrointestinal tract but are physically unable to manage nutritional intake through normal mastication and deglutition.
  Entarik Feeding Tube System:
  The Entarik Feeding Tube System is designed to aid qualified operators in the placement of the Entarik Feeding Tube (Entarik FT) into the stomach of patients requiring enteral feeding. The Entarik FT is equipped with sensors designed to provide information about the location of the tube tip relative to the stomach, thus assisting in reducing the incidence of misplacement during first positioning. The Entarik Monitor also monitors the feeding tube position continuously during the course of feeding and automatically and in real-time alerts of tube migration.
  Arms: Entarik
Device: Entarik Feeding Tube System without monitoring — Entarik Feeding Tube:
  The Entarik Feeding Tube is intended for the administration of nutrition, fluids and medications by the nasoenteric route for patients who have an intact gastrointestinal tract but are physically unable to manage nutritional intake through normal mastication and deglutition.
  Entarik Feeding Tube System:
  The Entarik Feeding Tube System will collect data from the Entarik Feeding Tube. There will be no monitoring or dislodgement alerts, and no placement guidance.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Entarik Feeding Tube System in an adult ICU patient population for the administration of nutrition, fluids and medications.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to swallow tabletsAt least 18 years old
* Able to provide informed consent or ability to have a legally authorized representative provide informed consent
* Adults in the ICU requiring an 8Fr, 10Fr, or 12Fr NG tube. The size of the feeding tube should be determined clinically, and the Entarik Feeding Tube should only be placed if that size is appropriate.
* Suitable to start enteral (gastric but no post-pyloric) feeding
* Anticipated to receive enteral feeding (either bolus or continuous feeds) for more than 6 hours and conclude the enteral nutrition while in the care of the ICU. If enteral nutrition has already been initiated, indicated for replacement of an NG feeding tube Note: Both subjects on a ventilator (non-invasive or invasive ventilation) or not requiring a ventilator are eligible for this study.

Exclusion Criteria:

* inability to receive a feeding tube including subjects with known history of issues such as esophagitis or strictures, frequent nose bleeds, basilar skull fracture or GI bleeding disorders
* Known major upper airway malformation
* Known major GI abnormality, upper GI malignancy, or partial gastric resection
* History of gastroparesis
* Currently pregnant
* NPO status - expected to remain NPO for the following 72 hours.
* Patient needs an MRI in the immediate future (e.g., 6-12h) where placement of the feeding tube (non-MRI compatible) is going to mandate replacement with standard feeding tube
* Critically ill, facing imminent death
* Deemed unsuitable for enrollment in study by the investigator based on subject's history (e.g., active anticoagulation therapy) or physical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Percentage of accurate verifications of anatomical locations of the tip of the Entarik feeding tube. The position of the feeding tube tip as processed by the Entarik placement algorithm will be compared to x-ray. | 1 year
  All patients will receive placement verification per institutional standard of care.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nova Clinical Research at HCA Florida Blake Hospital, Bradenton, Florida
  - HCA Chippenham and Johnston-Willis Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No